CLINICAL TRIAL: NCT00842660
Title: Phase III Trial for Primary Radiotherapy With Single-Agent Cisplatin or Combination Chemotherapy in PET/CT Defined Poor-Prognostic Cervical Cancer Patients
Brief Title: Radiotherapy With Single-Agent Cisplatin or Combination Chemotherapy in Defined Poor-Prognostic Cervical Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Department of Obstetrics & Gynecology, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 97-1165A3
Record Dates: First submitted 2009-02-08; First posted 2009-02-12 (Estimated); Last update posted 2010-01-05 (Estimated); Status verified 2009-02

CONDITIONS: Cervical Cancer
Keywords: Cervical cancer; concurrent chemoradiotherapy; gemcitabine
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemzar,survival (Experimental)
  Interventions: Drug: Gemzar (gemcitabine)

INTERVENTIONS:
Drug: Gemzar (gemcitabine) — Gemzar(gemcitabine) Hcl has 2'deoxy-2,2'-difluorouridine monohydrochloride
  Other Names: GEMCITABINE

SUMMARY:
Concurrent radiotherapy with cisplatin-based chemotherapy has become the standard treatment for patients with cervical cancer. However, in patients with advanced cervical cancer, half of them treated with contemporary radiotherapy plus single agent cisplatin still suffered from the local or distant relapse. How to improve the treatment outcome of these patients is a very important issue and requires further clinical investigation.

The major aim of this project is to conduct a prospective, randomized phase III clinical trial to examine if cervical cancer patients treated by radiotherapy with cisplatin and gemcitabine have better survival rates than those treated by radiotherapy with cisplatin alone.

Gemcitabine has been demonstrated to be a good radiosensitizer. In keeping with this, few clinical trials in early phases showed promising results when using concurrent radiotherapy with cisplatin and gemcitabine. According to these positive results, the investigators expect this trial has the potential to improve the survival in patients with advanced cervical cancer, reduce the medical costs due to tumor relapse, and then benefit the whole society.

DETAILED DESCRIPTION:
I). Study end points Primary end point: Patient survival, including overall survival and progression-free survival.

Secondary end points:

1. Acute toxicity during treatment
2. Tumor response rates
3. Sites of recurrence
4. Long-term complications and quality of life II). Design of study

An open-label, prospective randomized trial with two treatment arms:

* Arm I: Patients receive CCRT with weekly cisplatin only.
* Arm II: Patients receive CCRT with cisplatin plus gemcitabine. III). Study population 1) Number of subjects: A total of 172 patients (86 per treatment arm) will be accrued for this study within 4 years.

Conduct of study

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary squamous cell carcinoma of the uterine cervix.
* Previously untreated disease.
* Clinical FIGO stage III-IVa or pelvic/para-aortic lymph node positive by PET examination.
* No known metastases to supraclavicular nodes or other organs outside the radiotherapy field.
* Ages eligible: 35 years - 70 years.
* Patients must have adequate bone marrow, pulmonary, liver and renal function documented before radiotherapy. WBC > 3000/mm3, platelet > 100,000/mm3, serum transaminases (GOT, GPT) < 60 IU/ml, total bilirubin < 1.5mg%, creatinine < 1.4mg% (creatinine clearance > 60 ml/min).
* Performance status 0 or 1 (see Appendix I).
* The interval between RT and randomization is not greater than 3 weeks.
* Patients must have signed informed consent to participate this study.

Exclusion Criteria:

* Age > 70 or < 35
* Medical or psychological condition that would preclude treatment.
* Previous chemotherapy or pelvic RT.
* Small cell carcinoma, adenocarcinoma or adenosquamous carcinoma.
* Patient unreliable for treatment completion and follow-up.

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2009-02; Primary Completion 2012-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Patient survival, including overall survival and progression-free survival. | 2012,

SECONDARY OUTCOMES:
1) Acute toxicity during treatment 2) Tumor response rates 3) Sites of recurrence 4) Long-term complications and quality of life | 2013

CONTACTS AND LOCATIONS:
Overall Officials: Chun Chieh Wang, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (2):
- Taiwan (2):
  - Chong Jong Wang,, Kaohsiung City
  - Chien-Sheng Tsai, Keelung

REFERENCES:
- [Derived] Wang CC, Chou HH, Yang LY, Lin H, Liou WS, Tseng CW, Liu FY, Liou JD, Huang KG, Huang HJ, Huang EY, Chen CH, Chang TC, Chang CJ, Hong JH, Lai CH. A randomized trial comparing concurrent chemoradiotherapy with single-agent cisplatin versus cisplatin plus gemcitabine in patients with advanced cervical cancer: An Asian Gynecologic Oncology Group study. Gynecol Oncol. 2015 Jun;137(3):462-7. doi: 10.1016/j.ygyno.2015.03.046. Epub 2015 Mar 28. PMID 25827291